CLINICAL TRIAL: NCT00910754
Title: A QT/QTc and Multi-dose PK Study of Abiraterone Acetate (CB7630) Plus Prednisone in Patients With Metastatic Castration- Resistant Prostate Cancer
Brief Title: A QT/QTc and Multi-Dose Pharmacokinetic Study of Abiraterone Acetate Plus Prednisone in Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016942; COU-AA-006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Prostate Neoplasms
Keywords: Prostate neoplasms; Metastatic castration resistant prostate cancer; Abiraterone acetate; CB7630
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abiraterone acetate (Experimental): Patients will take 1000 mg of abiraterone acetate once daily plus prednisone 5 mg twice daily orally (by mouth) until disease progression.
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone acetate — Abiraterone acetate 1000 mg (4 x 250 mg tablets) administered orally once daily.
Drug: Prednisone — Prednisone 5 mg tablets administered orally twice daily.

SUMMARY:
The purpose of this study is to determine the effect of abiraterone acetate plus prednisone on the conduction of electric charges within the heart and to determine the blood levels of abiraterone acetate following administration in patients with metastatic castration-resistant prostate cancer.

DETAILED DESCRIPTION:
This is an open-label (identity of assigned study drugs will be known) study to evaluate the effects of abiraterone acetate plus prednisone on the conduction of electric charges within the heart in male patients diagnosed with metastatic castration-resistant prostate cancer (a progressive form of prostate cancer that spreads to other parts of the body). At various time points outline in the protocol from Day -1 of Cycle 1 up to Day 2 of Cycle 2, patients will have electrocardiograms extracted from a 24 hour holter-monitor to evaluate the electrical activity of their heart. Efficacy will be assessed according to Prostate Cancer Working Group 2 and modified Response Evaluation Criteria In Solid Tumors criteria. Serial blood samples for pharmacokinetic analysis (how the drug concentrations change over time) will be collected and safety will be monitored throughout the study. Patients will take 1000 mg of abiraterone acetate once daily plus prednisone 5 mg twice daily orally (by mouth) until disease progression and will be followed up for up to 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell histology
* Documented metastatic disease
* Has not received chemotherapy or has no more than one line of cytotoxic chemotherapy or biologic therapy for treatment of castration resistant prostate cancer (CRPC)
* Documented prostate specific antigen (PSA) progression as assessed by the investigator according to Prostate Cancer Working Group 2 (PCWG2) criteria despite medical or surgical castration, or prostate cancer progression documented by radiographic progression according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria
* Surgically or medically castrated with testosterone levels of <50 ng/dL (<2.0 nM)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of <= 1
* Agrees to protocol-defined use of effective contraception
* Protocol-specified laboratory parameters

Exclusion Criteria:

* Serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection
* Abnormal liver function
* Uncontrolled hypertension
* Active or symptomatic viral hepatitis or chronic liver disease
* Known brain metastasis
* History of pituitary or adrenal dysfunction
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class II-IV heart disease or cardiac ejection fraction measurement of < 50 % at baseline
* Diagnosis of cardiac arrhythmia
* Treatment with anti-arrhythmic drugs primarily for cardiac arrhythmia
* Abnormal electrocardiogram
* Other malignancy (except non-melanoma skin cancer, that is active or has a ≥ 30% probability of recurrence within 24 months) History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug
* Surgery or local prostatic intervention within 30 days of the first dose
* Radiotherapy or immunotherapy within 30 days, or single fraction of palliative radiotherapy within 14 days of administration of Cycle 1 Day 1
* Any acute toxicities due to prior therapy that have not resolved to a NCI CTCAE (version 3.0) grade of <=1
* More than one prior cytotoxic chemotherapy or biologic therapy for treatment of CRPC
* Prior chemotherapy with mitoxantrone or other anthracyclines (ie, doxorubicin, daunomycin, epirubicin and idarubicin)
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of Cycle 1 Day 1
* Prior flutamide (Eulexin) treatment within 4 weeks of Cycle 1 Day 1
* Prior bicalutamide (Casodex), nilutamide (Nilandron, Anandron) within 6 weeks of Cycle 1 Day 1
* Previous abiraterone acetate or other investigational CYP17 inhibitor (eg, TAK-700)
* Previous investigational antiandrogens (eg, MDV3100, BMS-641988)
* Patients receiving anti-coagulant therapy
* Condition or situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with patient's participation in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-05; Primary Completion 2009-11 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Mean maximal change in electrocardiogram QTc | Baseline on Day -1 of Cycle 1 compared with Day 1 of Cycle 1, Cycle 2, Cycle 4 and every third cycle thereafter

SECONDARY OUTCOMES:
Number of participants with change from baseline electrocardiogram QTc >30 msec | Pre-dose Cycles 1, 2, 4, and every third cycle after Cycle 4, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose, and end of study visit (4 weeks after last dose of study drug)
Number of participants with change from baseline electrocardiogram QTc >60 msec | Pre-dose Cycles 1, 2, 4, and every third cycle after Cycle 4, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose, and end of study visit (4 weeks after last dose of study drug)
Number of participants affected by an adverse event | Up to 30 days after the last dose of study medication
Number of participants with change in cortrosyn stimulation test | Baseline and end of study visit (4 weeks after last dose of study drug)
Number of participants with change in serum blood levels of testosterone | Baseline and end of study visit (4 weeks after last dose of study drug)
Number of participants with change in adrenocorticotropic hormone | Baseline and end of study visit (4 weeks after last dose of study drug)
Mean plasma concentrations of abiraterone | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Maximum plasma concentrations of abiraterone | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Time to reach the maximum plasma concentration of abiraterone | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Area under the plasma-concentration-time curve from time 0 to the last quantifiable concentration of abiraterone | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Area under the plasma-concentration-time curve from time 0 to infinite time of abiraterone | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Elimination half-life of abiraterone | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Radiographic progression free survival | Up to Month 60
Overall survival | Up to Month 60
Number of participants with prostate specific antigen response | Week 12
Time to prostate specific antigen progression according to Prostate Cancer Working Group 2 criteria | Up to Month 60
Number of participants with objective radiographic response according to Prostate Cancer Working Group 2 criteria | Up to Month 60

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (8):
- United States (6):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Buffalo, New York
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Myrtle Beach, South Carolina
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - San Antonio, Texas
- Canada (2):
  - BC Cancer Agency-Vancouver, Vancouver, British Columbia
  - Vancouver, British Columbia

REFERENCES:
- See also: A QT/QTc and Multi-dose PK Study of Abiraterone Acetate (CB7630) Plus Prednisone in Patients with Metastatic Castration- Resistant Prostate Cancer — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=2396&filename=CR016942_CSR.pdf